CLINICAL TRIAL: NCT05697705
Title: Real-world Effectiveness oF the OxfoRd-astrazeneca Covid-19 Vaccine as a Second bOoster Dose in Brazil (REFORCO-BRAZIL)
Brief Title: Effectiveness of the Oxford-AstraZeneca COVID-19 Vaccine as a 2nd Booster, the REFORCO-Brazil Study
Acronym: REFORCO-B
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111R00028
Record Dates: First submitted 2023-01-23; First posted 2023-01-26 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
Keywords: COVID-19, Real-World Effectiveness, ChAdOx1 nCOV-19 vaccine, Second booster dose
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19; BNT162 Vaccine; Ad26COVS1; sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Population A: For evaluating second booster doses
  Interventions: Other: ChAdOx1 nCOV-19 vaccine (Vaxzeria); Other: BNT162b2 (Pfizer); Other: Ad26.COV2.S (Janssen); Other: CoronaVac (Sinovac)
- Population B: For evaluating first booster doses
  Interventions: Other: ChAdOx1 nCOV-19 vaccine (Vaxzeria); Other: BNT162b2 (Pfizer); Other: Ad26.COV2.S (Janssen); Other: CoronaVac (Sinovac)

INTERVENTIONS:
Other: ChAdOx1 nCOV-19 vaccine (Vaxzeria) — Used as 2nd booster, 1st booster, or primary series
Other: BNT162b2 (Pfizer) — Used as 2nd booster, 1st booster, or primary series.
Other: Ad26.COV2.S (Janssen) — Used as 2nd booster, 1st booster, or primary series.
Other: CoronaVac (Sinovac) — Used as 2nd booster, 1st booster, or primary series.

SUMMARY:
This study will address specific questions concerning the additional protection of the AZ COVID-19 vaccine as a second booster dose in preventing severe COVID-19 outcomes (hospitalisation, ICU admission etc) and will provide data to inform COVID-19 vaccine booster dose recommendations.

DETAILED DESCRIPTION:
In Brazil, second COVID-19 boosters became available to specific risk groups in early 2022. By June 2022, immunocompromised individuals aged 12 years and above, individuals aged 50 years and above, and healthcare workers were eligible for a second booster. The vaccines available for second booster doses in Brazil are produced by AstraZeneca (AZ), Janssen, Pfizer and Sinovac.

While several studies have estimated absolute vaccine effectiveness (aVE) or relative vaccine effectiveness (rVE) of second boosters of mRNA COVID-19 vaccines, only a single study has, to date, estimated aVE of AZ vaccine as a second booster dose, and no studies have estimated rVE for AZ vaccine as a second booster dose. As the pandemic progresses, more individuals are choosing to become vaccinated (and boosted) against COVID-19 and thus there is greater need to evaluate the additional protection offered by a second booster dose amongst individuals previously administered a first booster. This is particularly important in the context of waning protection of a first booster dose.

The primary objective is to estimate relative vaccine effectiveness (rVE) against COVID-19 hospitalization of the AZ COVID-19 vaccine as a second booster dose relative to a first booster dose only, of any COVID-19 vaccine, administered at least four months ago.

This study will also evaluate rVE of other vaccines used in Brazil as a second booster doses. The study will further evaluate rVE of all vaccines (including the AZ-COVID-19 vaccine) as a first booster dose relative to a complete primary series only, of any COVID-19 vaccine administered at least four months ago."

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for SARS between 01 January 2022 and 31 December 2022 (Population A) or hospitalised for SARS between 01 August 2021 and 31 December 2022 (Population B).
* Eligible for a second COVID-19 vaccine booster dose at the time of SARS hospitalization (i.e., aged 50+ or aged 18+ and either a HCW or with an IC) for second booster objectives [Population A] OR eligible for a first COVID-19 vaccine booster dose at the time of SARS hospitalisation (i.e., aged 18+) for first booster objectives [Population B].
* Results available for a RT-PCR and/or antigen test for SARS-CoV-2 conducted on a sample taken up to 14 days after symptom onset.
* Individuals have required matching variables (e.g. age and sex).

Exclusion Criteria:

* Hospitalized for COVID-19 within 3 months prior to date of current hospital admission for SARS
* Nosocomially-acquired infection (where SARS case is flagged as nosocomial and/or where symptom onset date is after hospitalisation date)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population A is for evaluating second booster doses and will consist of individuals aged 18 years and over with immunocompromising conditions, healthcare workers aged 18 years and over, and individuals aged 50 years and over.
  Population B is for evaluating first booster doses and will consist of all individuals aged 18 and over.
Sampling Method: Non-Probability Sample
Enrollment: 188814085 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
COVID-19 confirmed by a positive antigen test or RT-PCR test in an individual hospitalized for SARS | Sample date within 14 days prior to and up to 2 days after hospitalization.
  Study includes SARS hospitalizations between August 2021 and December 2022 for evaluation of 1st booster dose effectiveness, and SARS hospitalizations between January 2022 and December 2022 for evaluation of 2nd booster dose effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Techtrials Pesquisa e Tecnologia Ltda., São Paulo, Brazil

REFERENCES:
- [Derived] Meeraus W, Postema A, Gray CM, Lee A, Maria AS, Furtado BE, Conde-Sousa E, Ouwens M, Valverde DA, da Cunha CA, Barbosa AN, Corte C, Taylor S. Second booster doses of adenoviral- and mRNA-based COVID-19 vaccines increase protection against COVID-19 hospitalization: Final analysis from the REFORCO-Brazil real-world effectiveness study during Omicron. Vaccine. 2025 Apr 19;53:126955. doi: 10.1016/j.vaccine.2025.126955. Epub 2025 Mar 10. PMID 40068393
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00028&attachmentIdentifier=942e6628-8511-452b-aa3f-52e918459021&fileName=Clinical_Study_Report_(CSR)_Synopsis_RIMS_REEFORCO_for_CTT.pdf&versionIdentifier=